CLINICAL TRIAL: NCT04943640
Title: The Additional Effect of Different Taping Applications on Pain, Functionality, and Tissue Temperature in Patients With Lumbar Radiculopathy: A Randomized Controlled Study
Brief Title: The Additional Effect of Different Taping Applications in Patients With Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA18/340
Record Dates: First submitted 2021-06-12; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Low Back Pain, Recurrent; Kinesiotape; Quality of Life; Physiotherapy
Keywords: low back pain; kinesiotape; quality of life; skin temperature; physiotherapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- kinesio taping (Experimental): The patient was advised to clean the skin with alcohol and shave the hairy areas. The standing patient was asked to take off high heels if he/she was wearing them.
  The paravertebral technique was used with 5 cm x 5 m kinesio tape material. While the patient was standing in an upright position, two longitudinal pieces were cut by taking the tape and slightly rolling its corners. The patient was asked to lean forward. The lower end of the tape was attached 7 cm below the sacroiliac joint at the level of the paravertebral muscles and the patient was bent forward. The patient was asked to do a slight rotation to the left, and while in this position, the tape was attached to T11-T12 without stretching at all. Kinesio tape was attached to the opposite side of the vertebrae with the same procedure.
  Interventions: Other: kinesio taping
- rigid taping (Experimental): The patient was asked to lean forward, and 5 cm x 5 m rigid tape material was used in the right paravertebral region. When bonding the tape, first, the lower end of the tape was attached 7 cm below the sacroiliac joint at the level of the paravertebral muscles and the patient was bent forward. Then, the patient was asked to do a slight rotation to the left, and while in this position, the hypoallergenic tape (beta fix) was applied with no tension [23]. Then, rigid tape was applied upward onto the paravertebral muscles. The left paravertebral region was taped with the same procedure as the right paravertebral region .
  Interventions: Other: rigid taping
- placebo taping groups (Placebo Comparator): Placebo taping was applied to patients in this group using betafix, an elastic stabilization tape, as material. A straight line of betafix was applied to the non-painful scapular inferior alignment of the spine, right and left, while the patient was standing upright.
  Treatment with taping was administered to all groups every 2 days by the same physiotherapist .
  Interventions: Other: placebo taping

INTERVENTIONS:
Other: kinesio taping — Kinesio tape was developed by Kenzo Kase in the 1970s. It is an elastic tape, and its adhesive face is sinusoidal wavy. This feature has been shown to increase daily living activities and functions, as it supports the tissue while also allowing movement [12]. Kinesio tape lifts the skin and subcutaneous soft tissues of the fascia, which are painful and inflamed regions upon contractions seen in the tissue after tense adhesion to the skin. Therefore, it has been reported to reduce oedema and inflammation by creating more space and providing blood and lymphatic fluid flow.
  Arms: kinesio taping
Other: rigid taping — The tape material used in rigid (athletic) tape application is hard. It is used to position and unite the soft tissue, to protect the tissue from impact and to prevent local swelling.There are studies in the literature supporting the sensorimotor and proprioceptive sensation-enhancing effect of the athletic band, which provides a very good sensory input through the skin.
  Arms: rigid taping
Other: placebo taping — Placebo taping was applied to the patients in this group, using betafix, an elastic fixation band, as the material. The patient was told that taping would be applied. A straight line betafix was applied to the non-painful scapular inferior level of the spine on the right and left sides of the standing patient.
  Arms: placebo taping groups

SUMMARY:
Our study aims to compare the therapeutic effects of different taping materials and techniques on pain, functionality, and tissue temperature in patients with lumbar radiculopathy.

DETAILED DESCRIPTION:
Pain occurs due to the intervertebral disc; ligaments in the region; or degeneration, strain, and sprains in the muscles, neurogenic, inflammatory, infectious, or neoplastic problems caused by structures in and around the spine . Low back pain is a serious health problem, with a lifetime prevalence of 84% . According to the American Society of Pain's clinical practice guidelines, low back pain is classified into three categories: nonspecific low back pain, radiculopathy-induced low back pain, and low back pain associated with another specific cause. A multidisciplinary approach is recommended for the treatment of low back pain. Before pharmacological treatments, cognitive behavioral therapy, physiotherapy exercise programmes, electrical physical therapy modalities, manual therapy, and psychological therapy are frequently referenced treatment options. Taping is one of the conservative physical therapy methods that is often a preferred treatment in clinics. Rigid (athletic) taping and kinesiological taping are the most preferred taping techniques . Non-elastic taping material is used in the rigid taping application. It is used to position soft tissue and ensure that the tissues come together, are protected from contact, create compression, and prevent local swelling. Studies supporting the sensorimotor and proprioceptive sensory enhancing effects of rigid tape, which provides very good sensory input over the skin, are found in previous studies [7-9]. Unlike rigid tape, kinesio tape can be stretched up to 140% of its resting length due to its structure, which is the approximate stretching capacity of normal skin .

Although there are various studies related to this topic, there is still no consensus on the effectiveness of taping in patients with low back pain who have disc degeneration. The reason for this is that some studies show the positive effect of kinesio taping on the reduction of low back pain, but some cannot show the effect of taping or find any changes . The healing mechanisms of different taping treatments have not been fully clarified. Moreover, local temperature, which is one of the indicators of vascularization and tissue healing, has not been investigated widely. Our study aims to examine the effects of different taping materials and techniques on pain, functionality, and local tissue temperature in patients with lumbar radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* The criterion for inclusion in the study for volunteers was low back pain due to lumbar radiculopathy.

Exclusion Criteria:

* Exclusion criteria were skin disease, central nervous system damage, tumour in the spine, surgical operation of the spine, pregnancy, and rheumatic disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change from Roland-Morris Disability Questionnaire score at five weeks | before and after five weeks of treatment (10 sessions)
  The Roland-Morris Disability Questionnaire is a 24-item survey designed to assess the degree of functional limitation in patients with low back pain. The questionnaire answers are Yes-No (Yes: 1 point, No: 0 points), and high scores indicate severe disability
Change from Tissue temperature at five weeks | before and after five weeks of treatment (10 sessions)
  Regional tissue temperature was measured by digital electronic infrared thermography (FLIR-e63900, Wilsonville, OR, USA). This method is a non-invasive assessment tool that does not require intervention by the investigator. The investigator can see changes in the skin surface temperature of the patient and, the thermal differences of the measured point are shown on the monitor.

SECONDARY OUTCOMES:
Change from The Oswestry Low Pain Disability Questionnaire score at five weeks | before and after five weeks of treatment (10 sessions)
  The Oswestry Disability Index measures the degree to which low back pain affects the daily life activities of patients in 10 different aspects (severity of pain, personal care, lifting, walking, sitting, standing, sleeping, degree of change of pain, social life, and travel). There are six expressions under each item that mark what is appropriate for the patient's condition. The first phrase is scored as "0", and the sixth phrase as "5"; 0-4 points is considered no disability, 5-14 points light disability, 15-24 points medium disability, 25-34 points serious disability, and 35-50 points total functional disability. The minimum score taken from the scale is 0, and the maximum score is 50. Fifty points indicate the highest level of functional inadequacy .
Change from Pain severity at five weeks | before and after each session( five weeks of treatmant)
  The Visual Analogue Scale (VAS) was used to evaluate the severity of pain felt during the activities and rest of patients. The scale is horizontal in the form of a line 10 cm long, starting with "no pain" and ending with "excruciating pain". The pain was measured and recorded as "cm" between the point marked with no onset .

CONTACTS AND LOCATIONS:
Overall Officials: Tugce Bozkurt, Principal Investigator — Ufuk University; Rabia Tugba Kilic, Study Director — Ankara Yildirim Beyazıt University; Hayri Baran Yosmaoğlu, Study Chair — Baskent University
Locations (3):
- Turkey (Türkiye) (3):
  - Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Ankara
  - Departmant of Health Services Vocational School, Physical Thraphy and Rehablitation, Ufuk University, Ankara
  - Faculty of Health Sciences, Departmant of Physiotherapy and Rehabilitation, Baskent University, Ankara

REFERENCES:
- [Background] Silva Parreira Pdo C, Menezes Costa Lda C, Takahashi R, Hespanhol Junior LC, Motta Silva T, da Luz Junior MA, Pena Costa LO. Do convolutions in Kinesio Taping matter? Comparison of two Kinesio Taping approaches in patients with chronic non-specific low back pain: protocol of a randomised trial. J Physiother. 2013 Mar;59(1):52; discussion 52. doi: 10.1016/S1836-9553(13)70147-4. PMID 23419916
- [Background] Yakut E, Duger T, Oksuz C, Yorukan S, Ureten K, Turan D, Frat T, Kiraz S, Krd N, Kayhan H, Yakut Y, Guler C. Validation of the Turkish version of the Oswestry Disability Index for patients with low back pain. Spine (Phila Pa 1976). 2004 Mar 1;29(5):581-5; discussion 585. doi: 10.1097/01.brs.0000113869.13209.03. PMID 15129077
- [Background] Kucukdeveci AA, Tennant A, Elhan AH, Niyazoglu H. Validation of the Turkish version of the Roland-Morris Disability Questionnaire for use in low back pain. Spine (Phila Pa 1976). 2001 Dec 15;26(24):2738-43. doi: 10.1097/00007632-200112150-00024. PMID 11740366
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Xue EY, Chandler LK, Viviano SL, Keith JD. Use of FLIR ONE Smartphone Thermography in Burn Wound Assessment. Ann Plast Surg. 2018 Apr;80(4 Suppl 4):S236-S238. doi: 10.1097/SAP.0000000000001363. PMID 29489530